CLINICAL TRIAL: NCT04547803
Title: Post-discharge Early Assessment With Remote Video Link (PEARL) Initiative: A Randomized Controlled Trial
Brief Title: Post-discharge Early Assessment With a Video-visit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sagar Dugani, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-004688
Record Dates: First submitted 2020-09-08; First posted 2020-09-14 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Hospital Discharge
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video Visit and Standard of Care (Experimental): Participants will participate in a video visit and standard of care
  Interventions: Other: Standard of Care; Other: Video Visit
- Standard of Care (Active Comparator): Participants will participate in standard of care for discharged patients.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Standard of Care — Outpatient appointments and activities including radiologic procedures for discharging patients as standard of practice
Other: Video Visit — 15-20 minute Video visit with an advanced practice provider (nurse practitioner or physician assistant) approximately 2-5 days after discharge.
  Arms: Video Visit and Standard of Care

SUMMARY:
The purpose of this study is to determine if a video visit with an advanced practice provider (Nurse Practitioner or Physician Assistant) within 7 days of discharge from Hospital Internal Medicine services will increase patient compliance with medication, self-management and home supports after hospital discharge.

DETAILED DESCRIPTION:
Prior to discharge, patients will be referred by Hospital Internal Medicine (HIM) teams to the PEARL team and screened for study eligibility. Eligible patients who provide oral consent to participate. Participants will be randomized 1:1 with comparisons between "Usual care" and "Usual care + Video-visit" arms. Participants randomized to the intervention arm will participate in a 15-20 minute Video visit (using Zoom®) with an advanced practice provider (APP; nurse practitioner or physician assistant in HIM) approximately 2-5 days after discharge. The telephone follow-up will occur 3-6 days after discharge. If a patient has a Video visit, the telephone follow-up will be scheduled for after the Video visit.

It is standard practice for HIM teams to make and coordinate outpatient appointments and activities including radiologic procedures for discharging patients. During this study, usual care will continue for patients in each arm. The intervention (Video-visit) is in addition to and not in place of the usual standard of care.

If issues/concerns beyond the scope of the video visit or telephone follow-up arise, then the PEARL APP will direct these to the discharging hospitalist team/supervising physician, or the participant's primary care provider (PCP) consistent with current standards of practice and management of post-discharge issues. Issues re-directed to the discharging hospitalist team or other providers will be documented in the Video-visit encounter. If the APP deems the clinical situation urgent or emergent, the APP will refer the patient to emergency services, or if needed ask the patient his/her location and contact 911. The APP will also immediately notify the study PI or co-PI who are both hospitalists and familiar with the practice. The APP will also notify the discharging hospitalist team.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years
* Patients discharged from a Hospital Internal Medicine service at Saint Marys Hospital
* Patients or their legally authorized representative provides consent to participate in the study
* Patients discharged home or to assisted living facility

Exclusion Criteria:

* Patients discharged from Hospital Service Meds 1-4 and Med 17
* Patient discharged with Care Transitions Program, or to Hospice, skilled nursing facility (SNF) or long-term acute care (LTAC) facility
* Post-procedure patients (i.e., elective hospital admission for planned intervention or procedure)
* Patient/legally authorized representative is Non-English speaking
* Patient leaves the hospital Against Medical Advice (AMA)
* No access to mobile technology/laptop/computer for post-discharge follow-up
* Patient with an active diagnosis Covid-19 infection
* Patients with a scheduled re-admission for a procedure, chemotherapy, or other treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1190 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Adherence to post-discharge recommendations | Through study completion, approximately 30 days
  Number of participants to adhere to post-discharge recommendation including medication compliance, self-management, and home supports post hospital discharge

SECONDARY OUTCOMES:
7 day readmission rate | 7 days after hospital discharge
  Number of participants with hospital emergency department visits and hospital readmission within 7 days of discharge
30 day readmission rate | 30 days after hospital discharge
  Number of participants with hospital emergency department visits and hospital readmission within 30 days of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Chandrasagar (Sagar) Dugani, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dugani SB, Kiliaki SA, Nielsen ML, Fischer KM, Lunde M, Kesselring GM, Lawson DK, Coons TJ, Schenzel HA, Parikh RS, Pagali SR, Liwonjo A, Croghan IT, Schroeder DR, Burton MC. Postdischarge Video Visits for Adherence to Hospital Discharge Recommendations: A Randomized Clinical Trial. Mayo Clin Proc Digit Health. 2023 Sep;1(3):368-378. doi: 10.1016/j.mcpdig.2023.06.006. Epub 2023 Aug 4. PMID 37641718
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials